CLINICAL TRIAL: NCT02531464
Title: Effectiveness of a Multi-faceted Intervention to Improve Supportive Care for Family Caregivers of Patients With Lung Cancer
Brief Title: Intervention to Improve Supportive Care for Family Caregivers of Patients With Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FRQS-30740
Record Dates: First submitted 2015-07-15; First posted 2015-08-24 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Lung Cancer
Keywords: family caregiver; quality of life; supportive care; distress screening; needs assessment
MeSH Terms: conditions — Lung Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: supportive care (Experimental): Family caregivers (FC) in the experimental arm (supportive care) will be exposed to a multi-faceted intervention to help them cope with their caregiving role, support them and respond to their needs; the intervention includes 3 components: 1) systematic distress screening and problems assessment of FCs at 2-month interval during the study period; 2) privileged contact with an oncology nurse away from the patient to further identify and address FCs' problems; 3) liaison by the oncology nurse with the family physician of FCs fwho will have reported high distress or needing help
  Interventions: Other: Supportive care
- Control: usual care (No Intervention): In the control arm (usual care), FCs will assist to their relative initial visit to the pivot nurse in oncology (PNO) . The PNO screens patients for distress and assesses their needs. She does a bio-psycho-social comprehensive evaluation and may provide help and information. She responds to questions and refers to appropriate resources, staying available for patients and their FCs throughout the cancer care trajectory. However, most PNO interventions target the patient, with no systematic distress screening and problems assessment for FCs, nor any service and resource specifically dedicated to them. If FCs clearly express distress or particular needs, the PNO will address them or refer to appropriate resources, but, in usual care, only few FCs receive support services

INTERVENTIONS:
Other: Supportive care — Systematic distress screening and needs assessment of family caregivers of patients with lung cancer
  Arms: Experimental: supportive care

SUMMARY:
Family caregivers play a crucial role in cancer patients care, as they are their principal source of support. It is well recommended to provide them with the resources, information and support needed to maintain a good health, and to sustain their caregiving role. Recently, oncology centres have implemented systematic distress screening programs, but the focus has been limited to cancer patients, with little intervention on family caregivers. This study aims to address this gap. It will implement and test the effectiveness of a simple intervention integrating primary care and oncology care that transfers into practice the main recommendations of governmental authorities and experts to globally improve supportive care. The intervention includes systematic distress screening and problems assessment of family caregivers at diagnosis, and every two months, privileged contact with a nurse away from the patient to address caregivers distress and identified problems, and for caregivers experiencing high level of distress, liaison by the study nurse with their family physician to transfer information on their identified problems and level of distress and to facilitate shared follow-up. This intervention has been pilot-tested with family caregivers, health care providers and decision makers involved in lung cancer care, as well as with community-based family physicians, to ensure its feasibility and acceptability. This study findings may clearly improve patient and caregiver experience of cancer care, and reduce the burden of disease.

DETAILED DESCRIPTION:
Lung cancer may cause severe distress not only in patients but also in their family caregivers (FCs), with a direct impact on quality of life (QoL). Distress can be higher in FCs than in patients. Results from a recent study on continuity of cancer care conducted by the investigators support these findings, as a significantly larger proportion of FCs than patients reported high levels of anxiety and distress early after the diagnosis of lung cancer and this difference remained after 6 and 12 months. Several cancer centers have implemented systematic distress screening program during the care trajectory, but they target only patients without extending it to FCs. This study aims to implement and assess the effectiveness of a multi-faceted intervention to improve supportive care for FCs of patients with lung cancer.

Specific objectives:

1. To assess the effectiveness of the intervention on:

   1.1 Caregivers' outcomes: distress (primary outcome), anxiety, depression, QoL, needs, burden, perception of health, preparedness in caregiving, perceived social support 1.2 Patients' outcomes: distress, anxiety, depression, QoL, pain and other symptom relief 1.3 Care process outcomes: FCs and patients' utilization of services
2. To further document and describe:

2.1 In the experimental group: FCs perceived usefulness of the intervention and perceived effect on distress/QoL 2.2 In the oncology team: perceived usefulness of the intervention and perceived effect on their practice/organization of care Methods: An experimental design is used to test the intervention during 9 months in a pulmonary oncology clinic in Quebec City where a distress screening tool is implemented for cancer patients (but not for FCs). A total of 120 FCs of patients newly diagnosed with a non-surgical lung cancer, followed at the clinic have been randomly assigned to either the intervention (experimental group N=60) or to usual care (control group N=60). Considering a 20% withdrawal rate (due to death or severe deterioration of patients' condition), this sample size allows to detect a 33% difference in distress scores between the two groups, with an estimated baseline distress score (with the HADS) of 13.7±7 (range 0-42), a 5% alpha error and a power of 80%. The intervention comprises 3 components: 1) systematic distress screening and problems assessment of FCs at their relative's cancer diagnosis and then, every 2 months for a maximum of 9 months; 2) privileged contact with an oncology nurse away from the patient to further identify and address FCs' problems; 3) liaison by the oncology nurse with the family physician of FCs who have reported a high level of distress (score ≥ 4 on the distress thermometer, which indicates a need for intervention), or who have mentioned needing help. In both groups, outcomes related to FCs and to care processes are measured with validated tools at baseline and every 3 months, for a maximum of 9 months. Measures are taken at the same intervals with patients since their physical and mental health may influence FCs' distress. Individual interviews with 12 FCs are planned to assess the usefulness of the intervention and its effect on their QoL. Interviews with the pivot nurses in oncology will document their satisfaction regarding the intervention and its effect on their practice.

Relevance. This translational study aims to assess the effectiveness of an intervention that transfers into practice the main recommendations of governmental authorities and experts regarding integrated care to globally improve cancer supportive care. It has the potential to make a significant impact on the burden of disease for FCs and to improve their quality of care. If proven effective, the conditions of success of this intervention could be replicated in other settings and for other types of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Relative identified by patients diagnosed with inoperable lung cancer as their principal family caregiver; having a family physician

Exclusion Criteria:

* Cognitive disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the mean score of distress (Hospital Anxiety Depression Scale) | Baseline, after 3, 6 and 9 months
  Measured by the Hospital Anxiety Depression Scale (HADS)
Change in the mean score of distress (Psychological distress scale used in the Quebec Health Survey) | Baseline, after, 3, 6 and 9 months
  Measured by the Psychological distress scale used in the Quebec Health Survey

SECONDARY OUTCOMES:
Change in the preparedness for Caregiving (8-item validated instrument) | Baseline, after 3, 6 and 9 months
  8-item validated instrument measuring the perceived readiness for multiple domains of the caregiving role (providing physical care, emotional support, setting up in-home support services and dealing with the stress of caregiving); the scale varies from 0 to 4
Change in the caregiver's Burden Scale in End of Life Care | Baseline, after 3, 6 and 9 months
  16-item instrument validated with FCs who assist cancer patients in palliative care; the scale varies from 1 to 4
Change in the family caregiver needs (Home Caregiver Need Survey) | Baseline, after 3, 6 and 9 months
  Measured by the Home Caregiver Need Survey, a 25-item tool covering informational, practical, emotional and spiritual needs. For each need, FCs indicate, on a 0 to 4 scale, its perceived importance and how well it is satisfied
Change in the family caregiver quality of life ( City-of-Hope Quality of Life Scale-Family Version) | Baseline, after 3, 6 and 9 months
  Measured by the City-of-Hope Quality of Life Scale-Family Version, a 37-item validated instrument that assesses 4 quality of life domains (physical, psychological, social and spiritual), with questions using a 0-10 scale; only the 4 items related to the general assessment of each quality of life domain will be used
Variation in service and health care resource utilization | Baseline, after 3, 6 and 9 months
  FCs will report the number of visits to their family physician and to any other health/psychosocial professional, meetings to support groups, use of community resources (volunteer services, respite, help for housework, etc.), use of sick leave, and prescription of sleeping pills, anxiolytic or antidepressant medications

CONTACTS AND LOCATIONS:
Overall Officials: Michele Aubin, MD, PhD, Principal Investigator — Laval University
Locations (1):
- Institut universitaire de cardiologie et pneumologie de Québec (IUCPQ), Québec, Quebec, Canada

REFERENCES:
- [Derived] Aubin M, Vezina L, Verreault R, Simard S, Desbiens JF, Tremblay L, Dumont S, Fillion L, Dogba MJ, Gagnon P. Effectiveness of an intervention to improve supportive care for family caregivers of patients with lung cancer: study protocol for a randomized controlled trial. Trials. 2017 Jul 4;18(1):304. doi: 10.1186/s13063-017-2044-y. PMID 28676071